CLINICAL TRIAL: NCT04084145
Title: National Unified Renal Translation Research Enterprise - Chronic Kidney Disease
Acronym: NURTuRE-CKD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Kidney Cancer UK (Other); UK Renal Registry (Unknown); University of Bristol (Other); University of Birmingham (Other); University of Southampton (Other); University of Geneva, Switzerland (Other); National Institute for Health Research, United Kingdom (Other Government); UCB Pharma Ltd (Unknown); Evotec International GmbH (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 16091
Record Dates: First submitted 2019-03-05; First posted 2019-09-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, DNA, renal biopsy tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD: Chronic Kidney Disease stage 1 - 4 followed up in secondary care

SUMMARY:
Chronic Kidney Disease (CKD) affects around 10% of the adult population and is associated with an increased risk of heart attack, stroke and end stage kidney disease (ESKD). This study aims to better predict who is most likely to progress to ESKD using previously identified risk factors and novel biomarkers in blood and urine samples, along with kidney biopsy tissue. Resources can then be directed to those most at risk of disease progression and other associated conditions such as heart attack and stroke, while those at lower risk can be offered less frequent monitoring.

DETAILED DESCRIPTION:
3,000 participants will be recruited from nephrology clinics at multiple participating centres (planned to start with 11). 100 control participants (without CKD) will be recruited from among hospital staff members, people attending diabetes clinics and the general public via advertisements placed in the hospitals and in the press.

Study participants with CKD will participate in the study for 12 - 18 months of active follow-up. After that participants will be sent a questionnaire annually by post to assess quality of life (EQ-5D-5L) and health care resource utilisation during the previous year and the investigators will collect outcome data without the need for further study visits; this annual follow-up by questionnaire will continue for 14 years following their second study visit.

Study participants acting as normal controls will attend only a single study visit.

All participants will provide written informed consent prior to undergoing any interventions. After providing written informed consent participants will undergo the following assessments and study procedures:

Medical History: The following data will be collected by interview, questionnaire and examination of the participants' medical records.

* Socio-demographic: age, gender, ethnicity, first language, education status, marital status, employment, indices of multiple deprivation (IMD) score (derived from postcode of residence), smoking history, alcohol intake, dietary status (vegetarian/vegan)
* Medical: All previous illnesses with particular focus on CKD diagnosis, previous AKI, hypertension, diabetes, cardiovascular disease (CVD), atrial fibrillation, rheumatoid arthritis, thyroid disease, retinopathy (if diabetic), peripheral neuropathy (if diabetic). These will be used to calculate the Charleston Comorbidity Index.
* Family medical history: CVD before age 60 years, diabetes, CKD, ESKD.
* All current medication including over the counter preparations and supplements/herbal preparations.
* Vaccination status for influenza and pneumococcus
* Prior laboratory results, especially prior serum creatinine results to enable analysis of trend in eGFR.
* The above data will be recorded on a questionnaire that participants will be asked to complete at or prior to the baseline study visit. Questionnaires will be checked by research staff at the study visit and participants will be assisted in completing the questionnaires if required. Details of the medical history and blood results will be verified by inspection of participants' hospital medical records.Quality of Life and Functional Status
* Quality of life will be measured by EQ-5D-5L quality of life questionnaire
* Functional status will assessed using the Karnofsky score
* Current symptoms will be assessed using an Palliative Outcome Scale (POS) questionnaire (POS-Renal P7)
* Health literacy will be assessed by questionnaire (single question SILS)
* Cognitive function will be assessed with the "six item Cognitive Impairment Test" (6CIT) questionnaire
* Anxiety and depression symptoms will be assessed with the "Hospital Anxiety and Depression Scale" (HADS)

Anthropomorphic assessment:

* Height
* Weight
* Body Mass Index
* Hip to waist ratio
* Waist circumference
* Mid-upper arm muscle circumference
* Hand grip strength
* Blood pressure (seated; average of 3 readings recorded with an oscillometric device in accordance with British Hypertension Society guidelines)
* Urine dipstick test
* "Timed up and go" (TUG) test

Laboratory Assays:

The following tests to be performed as part of routine clinical care:

* Urea and electrolytes
* Estimated GFR
* Magnesium, calcium and phosphate
* Serum albumin
* Lipid profile (including triglycerides)
* Random blood glucose
* Haemoglobin A1C (if diabetic)
* Bicarbonate
* Uric acid
* Full blood count
* High sensitivity C-reactive protein (CRP)
* Ferritin (if anaemic)
* Folic acid (if anaemic)
* Vitamin B12 (if anaemic)
* Serum Parathyroid hormone
* Urine albumin to creatinine ratio
* Urine protein to creatinine ratio

Specimens for Biorepository: In addition to the routine biochemistry detailed above, additional biosamples will be obtained from each participant at each study visit as follows:

* 10ml plasma (30mL of blood)
* 10ml serum (30mL of blood)
* 2 x 3ml whole blood for DNA extraction: genomics and epigenetics
* 1 x 2,5ml whole blood for RNA extraction
* 100ml urine

Participants acting as controls will undergo the following assessments and study procedures after signing written informed consent:

Socio-Demographic data:

Participants will be asked to give their sex and date of birth as well as post code of residence (to derive indices of multiple deprivation score)

Anthropomorphic Assessment:

* Height
* Weight
* Body Mass Index
* Hip to waist ratio
* Waist circumference

Laboratory Assays:

* Urea and electrolytes
* Estimated GFR
* Urine albumin to creatinine ratio
* Random blood glucose
* High sensitivity C-reactive protein
* Haemoglobin A1C (if diabetic)

Specimens for Biorepository: In addition to the biochemistry detailed above, additional biosamples will be obtained as follows:

* 10ml plasma (30mL of blood)
* 10ml serum (30mL of blood)
* 100ml urine
* 2 x 3ml whole blood for DNA extraction: genomics and epigenetics
* 1 x 2,5ml whole blood for RNA extraction

Control participants will undertake a single study visit. Participants with CKD will undertake a study visit 2 12-18 months from the date of the first study visit. In addition participants will be asked to complete a health utilisation questionnaire to obtain details regarding hospital admissions, GP visits and medication changes during the year since recruitment Compliance will be defined by attendance at the second study visit.

Criteria for terminating trial The study will be discontinued only if for unforeseen circumstances it becomes clear that it is no longer feasible. If a participating centre is unable to recruit successfully, it will be withdrawn from the study and replaced by another centre. Participants already recruited from a centre that withdraws from the study will remain in the study.

ELIGIBILITY:
Participants with CKD

Inclusion Criteria:

1. Age Over 18 years of age
2. Estimated GFR 59-15ml/min/1.73m² or eGFR >60ml/min/1.73m² and urine albumin to creatinine ratio >30mg/mmol
3. Seen at least once in a Nephrology Clinic
4. Willing to participate in two study visits
5. Able to give informed consent and participate in study procedures

Exclusion Criteria:

1. Recipient of a solid organ transplant
2. Expected survival less than 1 year (in the opinion of local investigators)
3. Acute kidney injury within 3 months of recruitment
4. Major Acute Cardiovascular Event (MACE) within 3 months of recruitment

Participants without CKD - controls Inclusion criteria

1. Age over 18 years of age
2. Willing to participate in one study visit
3. Able to give informed consent and participate in study procedures
4. No evidence of CKD
5. No other major illnesses except for hypertension and type 2 diabetes mellitus (50 participants will have diabetes but no CKD)

Exclusion criteria

1. Estimated GFR<60ml/min/1.73m2 in previous 12 months or last available result
2. Urine albumin to creatinine ratio >3mg/mmol in previous 12 months or last available result
3. Previous unilateral nephrectomy or partial nephrectomy
4. Recipient of a solid organ transplant
5. Expected survival less than 1 year (in the opinion of local investigators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from nephrology clinics at multiple (planned to start with 11) participating sites.
  Control participants (without CKD) will be recruited from among hospital staff members, people attending diabetes clinics and the general public.
Sampling Method: Non-Probability Sample
Enrollment: 3004 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with CKD progression | 5 years
  Progression of chronic kidney disease to kidney failure (defined as sustained decrease to <15mL/min/1.73m2 or initiation of kidney replacement therapy).
Number of participants who experience a major acute cardiovascular event | 5 years
  Cardiac death, non-fatal myocardial infarction, cerebral infarction or intracerebral haemorrhage , arterial revascularisation

SECONDARY OUTCOMES:
Rate of GFR decline | 5 years
  Rate of GFR decline calculated from serial eGFR values
Rate of GFR decline | 10 years
  Rate of GFR decline calculated from serial eGFR values
Rate of GFR decline | 15 years
  Rate of GFR decline calculated from serial eGFR values
Number of participants with CKD progression | 5 years
  Progression of CKD as defined by a 50% , 40 % or 30% reduction in estimated eGFR
Number of participants with CKD progression | 10 years
  Progression of CKD as defined by a 50% , 40 % or 30% reduction in estimated eGFR
Number of participants who experience a major acute cardiovascular event | 15 years
  Cardiac death, non-fatal myocardial infarction, cerebral infarction or intracerebral haemorrhage
Number of participants who die from any cause | 5 years
  Death from any cause
Number of participants who die from any cause | 10 years
  Death from any cause
Number of participants who die from any cause | 15 years
  Death from any cause
Number of participants who progress to end stage kidney disease (ESKD) | 5 years
  Development of end stage kidney disease (ESKD = eGFR <15mL/min/1.73m2)
Number of participants who progress to end stage kidney disease (ESKD) | 10 years
  Development of end stage kidney disease (ESKD = eGFR <15mL/min/1.73m2)
Number of participants who progress to end stage kidney disease (ESKD) | 15 years
  Development of end stage kidney disease (ESKD = eGFR <15mL/min/1.73m2)
Number of participants who experience acute kidney injury (AKI) | 5 years
  Development of AKI (KDIGO definition)
Number of participants who experience acute kidney injury (AKI) | 10 years
  Development of AKI (KDIGO definition)
Number of participants who experience acute kidney injury (AKI) | 15 years
  Development of AKI (KDIGO definition)
Number of participants admitted to hospital with a new diagnosis of cardiac failure | 5 years
  Number of participants admitted to hospital with a new diagnosis of cardiac failure
Number of participants admitted to hospital with a new diagnosis of cardiac failure | 10 years
  Number of participants admitted to hospital with a new diagnosis of cardiac failure
Number of participants admitted to hospital with a new diagnosis of cardiac failure | 15 years
  Number of participants admitted to hospital with a new diagnosis of cardiac failure
Number of participants with an unplanned hospital admission | 5 years
  Number of participants with an unplanned hospital admission
Number of participants with an unplanned hospital admission | 10 years
  Number of participants with an unplanned hospital admission
Number of participants with an unplanned hospital admission | 15 years
  Number of participants with an unplanned hospital admission
Number of participants admitted to hospital with an infection | 5 years
  Number of participants admitted to hospital with an infection
Number of participants admitted to hospital with an infection | 10 years
  Number of participants admitted to hospital with an infection
Number of participants admitted to hospital with an infection | 15 years
  Number of participants admitted to hospital with an infection
Number of participants with a new diagnosis of cancer | 5 years
  Number of participants with a new diagnosis of cancer
Number of participants with a new diagnosis of cancer | 10 years
  Number of participants with a new diagnosis of cancer
Number of participants with a new diagnosis of cancer | 15 years
  Number of participants with a new diagnosis of cancer
Number of participants with a hip fracture | 5 years
  Number of participants with a hip fracture
Number of participants with a hip fracture | 10 years
  Number of participants with a hip fracture
Number of participants with a hip fracture | 15 years
  Number of participants with a hip fracture
Number of participants with progression of chronic kidney disease (CKD) (KDIGO definition) | 5 years
  Progression of CKD (KDIGO definition:25% reduction in GFR and progression to next CKD category)
Number of participants with progression of chronic kidney disease (CKD) (KDIGO definition) | 10 years
  Progression of CKD (KDIGO definition:25% reduction in GFR and progression to next CKD category)
Number of participants with progression of chronic kidney disease (CKD) (KDIGO definition) | 15 years
  Progression of CKD (KDIGO definition:25% reduction in GFR and progression to next CKD category)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Taal, MBChB, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Royal Derby Hospital, Derby, Derbyshire
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Yes
Application for use of data to the independent NURTuRE Steering Group, facilitated by Kidney Research UK
Supporting Information: Study Protocol, SAP, CSR
Time Frame: variable depending on applications
Access Criteria: Approval of application by independent NURTuRE Steering Group
URL: https://nurturebiobank.org

REFERENCES:
- [Result] Taal MW, Lucas B, Roderick P, Cockwell P, Wheeler DC, Saleem MA, Fraser SDS, Banks RE, Johnson T, Hale LJ, Andag U, Skroblin P, Bayerlova M, Unwin R, Vuilleumier N, Dusaulcy R, Robertson F, Colby E, Pitcher D, Braddon F, Benavente M, Davies E, Nation M, Kalra PA. Associations with age and glomerular filtration rate in a referred population with chronic kidney disease: methods and baseline data from a UK multicentre cohort study (NURTuRE-CKD). Nephrol Dial Transplant. 2023 Oct 31;38(11):2617-2626. doi: 10.1093/ndt/gfad110. PMID 37230953
- [Result] Phillips T, Harris S, Aiyegbusi OL, Lucas B, Benavente M, Roderick PJ, Cockwell P, Kalra PA, Wheeler DC, Taal MW, Fraser SDS. Potentially modifiable factors associated with health-related quality of life among people with chronic kidney disease: baseline findings from the National Unified Renal Translational Research Enterprise CKD (NURTuRE-CKD) cohort. Clin Kidney J. 2024 Jan 19;17(2):sfae010. doi: 10.1093/ckj/sfae010. eCollection 2024 Feb. PMID 38313684
- [Result] Lucas BJ, Cockwell P, Fraser SDS, Kalra PA, Wheeler DC, Taal MW. Associations With Baseline Blood Pressure Control in NURTuRE-CKD. Kidney Int Rep. 2024 Feb 15;9(5):1508-1512. doi: 10.1016/j.ekir.2024.02.013. eCollection 2024 May. No abstract available. PMID 38707802
- [Result] McDonnell T, Kalra PA, Vuilleumier N, Cockwell P, Wheeler DC, Fraser SDS, Banks RE, Taal MW. The Impact of Primary Renal Diagnosis on Prognosis and the Varying Predictive Power of Albuminuria in the NURTuRE-CKD Study. Am J Nephrol. 2025;56(1):1-12. doi: 10.1159/000541770. Epub 2024 Oct 4. PMID 39369692
- See also: study web page — https://nurturebiobank.org

DOCUMENTS (1):
  • Study Protocol (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04084145/Prot_001.pdf